CLINICAL TRIAL: NCT03868540
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Oral Doses of BI 1291583 qd Versus Placebo in Healthy Male and Female Subjects for 4 Weeks (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: A Study in Healthy Men and Women to Find Out How Well Different Doses of BI 1291583 Are Tolerated
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1397-0002; 2018-001245-14 (EudraCT Number)
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1291583 (Experimental)
  Interventions: Drug: BI 1291583
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1291583 — tablet
  Other Names: Verducatib
  Arms: BI 1291583
Drug: Placebo — tablet
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1291583 in healthy male and female subjects following oral administration of multiple rising doses over 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male, or female (of non-childbearing potential) subjects -- For 'female of non-childbearing potential' at least one of the following criteria must be fulfilled:

  * Permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy)
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with FSH above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR), or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking during in-house confinement
* Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with 'women of childbearing potential' (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after the last administration of trial medication
* Known relevant immunodeficiency
* History and/or presence of tuberculosis; positive result for interferon gamma release assay (IGRA) (i.e., QuantiFERON TB-Gold)
* Positive results for Hepatitis B antigen, Hepatitis C antibodies and/or human immunodeficiency virus (HIV) 1 antigen or HIV1/2 antibodies, at screening
* Aural body temperature of more than 37.7°C on Day -3 to -1
* Volunteers who have received live or live-attenuated vaccine in the 4 weeks prior to dosing
* C-reactive protein above upper limit of laboratory reference range at screening and/or on Day -3 to -1
* Subjects with signs of current gingivitis/periodontitis. Inspection of the oral cavity will be performed by the investigator
* Subjects with a history of hyperkeratosis or erythema in palms or soles

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with drug-related adverse events | From first intake of trial medication until 21 days (Residual Effect Period) after the last drug administration, up to 49 days.
  Percentage of participants with drug-related adverse events.

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose (AUCτ,1) | Within 3 hours (h) before the first drug administration and 1, 2, 4, 6, 8, 10, 12, 14, 24 hours afterwards.
  Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose (AUCτ,1).
Maximum measured concentration of the analyte in plasma after administration of the first dose (Cmax,1) | Within 3 hours (h) before the first drug administration and 1, 2, 4, 6, 8, 10, 12, 14, 24 hours afterwards.
  Maximum measured concentration of the analyte in plasma after administration of the first dose (Cmax,1).
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Within 15 minutes prior to last drug administration (timepoint of last drug administration: 648 hours after first drug administration) and 1, 2, 4, 6, 8, 10, 12, 14 and 24 hours after the last drug administration.
  Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss).
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Within 15 minutes prior to last drug administration (timepoint of last drug administration: 648 hours after first drug administration) and 1, 2, 4, 6, 8, 10, 12, 14 and 24 hours after last drug administration.
  Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss).

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing